CLINICAL TRIAL: NCT06461858
Title: Effects of Cuevas Medek Exercises on Trunk Control and Balance in Children With Down Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & 23/0773
Record Dates: First submitted 2024-06-12; First posted 2024-06-17 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Down Syndrome
Keywords: Down syndrome; ,Trunk Control; Balance; conventional therapy.; Cuevas Medek exercises
MeSH Terms: conditions — Down Syndrome | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- This group (Group A) will receive cuevas medek technique (exercise) (Experimental): The first group, known as the experimental group, group A, receives Cuevas Medek exercises once a week, for 45 minutes per session,for 6 weeks.
  Interventions: Other: cuevas medek technique (exercise)
- This group (Group B) will receive conventional therapy. (Active Comparator): this second group, group B, referred to as the conventional therapy group (Routine physical therapy), follows a regimen of conventional therapy once a week for 6 weeks for 20 mints.
  Interventions: Other: conventional therapy

INTERVENTIONS:
Other: cuevas medek technique (exercise) — The first group, known as the experimental group, group A, receives Cuevas Medek exercises once a week, for 45 minutes per session,for 6 weeks
  Arms: This group (Group A) will receive cuevas medek technique (exercise)
Other: conventional therapy — Group B, referred to as the conventional therapy group (Routine physical therapy), follows a regimen of conventional therapy once a week for 6 weeks for 20 mints.
  Arms: This group (Group B) will receive conventional therapy.

SUMMARY:
Down syndrome, a genetic condition caused by the presence of an extra copy of chromosome 21. This additional genetic material affects the normal development of the brain and body, leading to intellectual and developmental delays. Individuals with Down syndrome often have distinctive physical features, such as a flat facial profile, almond-shaped eyes, and a short neck. Down syndrome has three types include Trisomy 21 (95% cases, extra chromosome 21), Translocation (3-4%, extra part attached), and Mosaic (1-2%, mixture of normal and trisomic cells). Children with Down syndrome often face challenges in motor development, including issues with muscle tone and coordination. However, targeted interventions and exercises, such as those focused on trunk control and balance, can have positive impact. The significance of this study is that it will define that specific exercises will affect the trunk control and balance in children with down syndrome.

This will be a randomized clinical trial; data will be collected from Rising Sun Institute in Lahore. Study will be conducted on 32 patients. The study will include children with Down syndrome aged between 2- and 6-years old children. Patients have uncontrolled epilepsy, Surgical or other medical intervention not included in study. In our data collection, there are two distinct groups, having same baseline of trunk control and balance. The first group, known as the experimental group, group A, receives Cuevas Medek exercises three times a week, twice a day, for 45 minutes per session, in contrast, group B, referred to as the conventional therapy group (Routine physical therapy), follows a regimen of conventional therapy 2 times a week for 6 weeks for 20 mints. Variables will be measured by following measurement tools:1. Trunk control measured through TIS (trunk impairment scale) assesses Static Sitting Balance, Dynamic Sitting Balance, and Coordination. 2. Pediatric Clinical Test of Sensory Interaction for Balance (P-CTSIB) used to identify the balance impairments in pediatric populations. 3.Balance appraised with the Berg Balance Scale (PBS). Pre and post assessment of trunk control and balance perform by these tools.

DETAILED DESCRIPTION:
Cuevas Medek Exercises (CME) is a pediatric physiotherapy approach for children with developmental motor delay impacting the central nervous system. According to Ramon Cuevas the creator of the method, its main principle involves provoking novel automatic motor reactions using exercises against gravity with progressive distal holdings. The physiotherapy intervention was composed of 1-hour sessions once or twice per week, and daily home program exercises. In CME interventions, the exercises are repeated 3, 5, or 8 times, depending on the effectiveness and the quality of the expected reaction. The better the reaction, the more repetitions are done .Moreover, different and more challenging exercises should be performed to provoke the brain to react in a new way (1).

Down syndrome (Ds) is an autosomal disorder caused by the presence of an extra chromosome 21, also known as trisomy 21. Statistics vary, but it is estimated that over 200,000 people in the United States today have Ds (2). Ds causes a range of intellectual disabilities and developmental delays in motor skills. The lifespan of people with Ds has increased from an average of 12 years in the 1940s to 60 years now for people with Ds in high-income countries. Most adults with Ds lead a sedentary lifestyle; previous research reported that less than 10% of adults with Ds achieve the recommended amount of physical activity. Adults with Ds often experience cardiovascular issues and generally higher rates of obesity than their peers, and low aerobic capacity. In addition to lower cardiovascular function, individuals with Ds exhibit lower strength compared with other sedentary peers. In children with Down syndrome, dysfunction of stereognosis and decrease in motor skills are also related to hypotonia. Hypotonicity disrupts the feedback mechanism which enables the perception of the position of the body in space, and plays a role in the voluntary control of muscles, and as a result body posture and the quality of movement are affected (3).

Children with weakened axial muscle tone face various problems every day. One is maintaining a stable body posture, which limits their participation in activities and games with peers. The study aimed to assess balance parameters in children with weakened axial muscle tone. Disturbances in ADL and IADL may be caused, among other things, by reduced muscle tone. Children with weakened muscle tone often have problems with properly integrating stimuli because skeletal muscles (whose strength is weakened in these children) are involved in mobility, strength, and balance, enabling participation and performance of various activities. Previous studies have shown that low muscle mass and strength contribute to adverse health effects in childhood, such as increased risk of metabolic dysfunctions, cardiovascular diseases, reduction of bone minerals or poorer cognitive and motor performance in early childhood compared to other children of the same age. These children in the later period struggle not only with motor difficulties but also with cognitive ones. There are several neuromuscular and musculoskeletal characteristics in Down syndrome which can result in developmental delays, generalized hypotonia and laxity of the joints due to hypotonia are present (1).

These factors may cause motor and postural delays, sensory processing and sensory integration deficits due to limitations in primary sensory experiments. when the sensory and motor interventions are performed earlier, it is probably more effective on the improvement of generation of new synapses and prevention of decrease in synapses in the next years of the life of these children and more neuro-plasticity of the nervous system .Individuals with Ds often have significant involvement of the musculoskeletal system, including ligamentous laxity and low muscle tone , leading to a higher risk of pes planus, scoliosis, hip disorders, and patellar instability if untreated. Strengthening of core muscles and joint stabilizers are frequently recommended strategies to counteract the effects of ligamentous laxity and low muscle tone (2).

This study aims will investigate the impact of Cuevas Medek exercises on trunk control and balance in children with Down syndrome. Additionally, it seeks to discern any distinctions in outcomes between conventional exercises or strength training alone and a combination of conventional exercises and Cuevas Medek exercises in terms of trunk, abdominal, lumbar endurance, and overall balance in this specific population of children with down syndrome.

Down syndrome, a genetic condition caused by the presence of an extra copy of chromosome 21. This additional genetic material affects the normal development of the brain and body, leading to intellectual and developmental delays. Individuals with Down syndrome often have distinctive physical features, such as a flat facial profile, almond-shaped eyes, and a short neck. Down syndrome has three types include Trisomy 21 (95% cases, extra chromosome 21), Translocation (3-4%, extra part attached), and Mosaic (1-2%, mixture of normal and trisomic cells). Children with Down syndrome often face challenges in motor development, including issues with muscle tone and coordination. However, targeted interventions and exercises, such as those focused on trunk control and balance, can have positive impact. The significance of this study is that it will define that specific exercises will affect the trunk control and balance in children with down syndrome.

This will be a randomized clinical trial; data will be collected from Rising Sun Institute in Lahore. Study will be conducted on 32 patients. The study will include children with Down syndrome aged between 2- and 6-years old children. Patients have uncontrolled epilepsy, Surgical or other medical intervention not included in study. In our data collection, there are two distinct groups, having same baseline of trunk control and balance. The first group, known as the experimental group, group A, receives Cuevas Medek exercises three times a week, twice a day, for 45 minutes per session, in contrast, group B, referred to as the conventional therapy group (Routine physical therapy), follows a regimen of conventional therapy 2 times a week for 6 weeks for 20 mints. Variables will be measured by following measurement tools:1. Trunk control measured through TIS (trunk impairment scale) assesses Static Sitting Balance, Dynamic Sitting Balance, and Coordination. 2. Pediatric Clinical Test of Sensory Interaction for Balance (P-CTSIB) used to identify the balance impairments in pediatric populations. 3.Balance appraised with the Berg Balance Scale (PBS). Pre and post assessment of trunk control and balance perform by these tools

ELIGIBILITY:
Inclusion Criteria:

* All children with Ds between 2-6 years old children were eligible for inclusion (5).
* Encompass children with scores falling within 41-50 range on the Berg Balance Scale.
* Had not received any strengthening exercise program in past 3 months
* Consent from parents and participants should be taken.

Exclusion Criteria:

* Epilepsy
* Surgical or other medical intervention scheduled during the intervention period or up to three months prior to the trial
* Participant unable to give clear voluntary assent and/or no written consent given by parent or guardian (5).
* Orthopedic condition or medical problems that prevent children from participating in exercise (4).

Ages: 2 Years to 6 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2024-08-10 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Trunk Impairment Scale for Trunk Control | Baseline and 6th Week
  This scale assesses the control in trunk muscles. The static subscale investigates: (1) the ability of the subject to maintain a sitting position with feet supported; (2) the ability to maintain a sitting position while the legs are passively crossed, and (3) the ability to maintain a sitting position when the subject crosses the legs actively. Interpretation: For each item, a 2-, 3- or 4-point ordinal scale is used. On the static and dynamic sitting balance and coordination subscales the maximal scores that can be attained are 7, 10 and 6 points. The total score for TIS ranges between 0 for a minimal performance to 23 for a perfect performance. Reliability: Intra-observer and inter-observer reliability is high. Test/retest and interobserver reliability for the TIS total score (ICC) - 0.96 and 0.99, respectively. Validity:(construct validity) was 0.86, between the TIS and the Trunk Control Test (concurrent validity) 0.83 (6).
Pediatric Clinical Test of Sensory Interaction for Balance for balance | Baseline and 6th Week
  This scale is used to identify the balance impairments in pediatric populations. Patient completes 3 trials of each of the 6 conditions (with hands on hips): stand on firm surface eyes open, stand on firm surface eyes closed, stand on firm surface with conflict dome, stand on foam eyes open, stand on foam eyes closed, stand on foam with conflict dome. The patient then completes all 6 conditions in narrow base of support with malleoli touching and tandem stance. The best score of 2 trials for each condition is documented (higher time or least sway). Timing is stopped if the child makes a postural adjustment (moving hands, feet, or eyes) (7).Reliability: Interrater=.69-.90; test-retest=.45-.78.Validity: construct validity= .63-.68 (8).

CONTACTS AND LOCATIONS:
Overall Officials: Fareeha Kausar, PP-DPT, Study Chair — Riphah International University; Hafiza Sara wafa, MS-PPT, Principal Investigator — Riphah International University
Locations (1):
- Al-Qaim Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jacewicz J, Dziuba-Slonina A, Chwalczynska A. Assessment of Balance Parameters in Children with Weakened Axial Muscle Tone Undergoing Sensory Integration Therapy. Children (Basel). 2023 May 7;10(5):845. doi: 10.3390/children10050845. PMID 37238393
- [Background] Verheyden G, Nieuwboer A, Mertin J, Preger R, Kiekens C, De Weerdt W. The Trunk Impairment Scale: a new tool to measure motor impairment of the trunk after stroke. Clin Rehabil. 2004 May;18(3):326-34. doi: 10.1191/0269215504cr733oa. PMID 15137564
- [Background] de Oliveira GR, Fabris Vidal M. A normal motor development in congenital hydrocephalus after Cuevas Medek Exercises as early intervention: A case report. Clin Case Rep. 2020 Apr 27;8(7):1226-1229. doi: 10.1002/ccr3.2860. eCollection 2020 Jul. PMID 32695363
- [Background] Westcott SL, Crowe TK, Deitz JC, Richardson PK. Test-retest reliability of the pediatric clinical test of sensory interaction for balance (P-CTSIB). Physical & Occupational Therapy in Pediatrics. 1994;14(1):1-22.
- [Background] Crowe TK, Deitz JC, Richardson PK, Atwater SW. Interrater reliability of the pediatric clinical test of sensory interaction for balance. Physical & Occupational Therapy in Pediatrics. 1991;10(4):1-27.
- [Background] Franjoine MR, Darr N, Held SL, Kott K, Young BL. The performance of children developing typically on the pediatric balance scale. Pediatr Phys Ther. 2010 Winter;22(4):350-9. doi: 10.1097/PEP.0b013e3181f9d5eb. PMID 21068635
- [Background] Mitroi S. Stimulation of triple extension tone and orthostatic balance in the child with cerebral palsy through exercises specific to Medek method. Physical Education, Sport and Kinesiology Journal. 2016;1(43):48-51.